CLINICAL TRIAL: NCT05259904
Title: Study to Improve dEployment Related Asthma by Using L-citrulline Supplementation (SEALS)
Brief Title: Study to Improve Deployment Related Asthma by Using L-Citrulline Supplementation
Acronym: SEALS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Jewish Health (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 21-2804; W81XWH2110677 (Other Grant/Funding Number: Department of Defense/USAMRAA); 21-2804 (Other: COMIRB); E02466 (Other: USAMRDC ORP HRPO)
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Post Deployment Related Asthma; Asthma
MeSH Terms: conditions — Asthma | interventions — Citrulline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- L-citrulline (Experimental): L-citrulline with a dose of 15 g/day will be administered in powder form that is mixed with water and taken orally, continuously and daily for at least 7 weeks. Dispensed at Visits 0a/1. Washout period of 4 to 6 weeks and then enter crossover phase of an additional 7 weeks. Drug will be dispensed at Visit 4.
  Interventions: Drug: L-citrulline
- Matching Placebo (Placebo Comparator): Administered in powder form that is mixed with water and taken orally, continuously, and daily for at least 7 weeks. Dispensed at Visits 0a/. Washout period of 4 to 6 weeks and then enter crossover phase of an additional 7 weeks. Drug will be dispensed at Visit 4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-citrulline — 7 weeks of treatment with 15 g/day of orally administered (powder form mixed with water) L-citrulline
  Arms: L-citrulline
Drug: Placebo — 7 weeks of treatment with orally administered matching placebo (to 15 g/day of L-citrulline)
  Arms: Matching Placebo

SUMMARY:
Service men and women returning from deployment are significantly more likely to develop asthma and severe respiratory symptoms from airway obstruction. Why this happens is not well known, but exposure to diesel, burn pits, biomass smoke, and sandstorms are thought to play a role. Ultimately, patients with deployment related asthma develop a complex airway disease that does not respond well to standard asthma medications. Therefore, it is imperative that safe and affordable treatments that could improve quality of life and symptoms are studied.

It has been previously shown that adult patients with poorly controlled asthma have an abnormal regulation of an amino acid called L-arginine and airway nitric oxide (FeNO), a gaseous molecule normally produced in the airways of healthy people. In healthy people, nitric oxide is present in amounts that help keep the airways open. However, in some patients with asthma, nitric oxide and L-arginine are often low. The investigators' preliminary data in obese asthmatics show that L-citrulline, which is an amino acid that can be metabolized into L-arginine, improved lung function and asthma control, while increasing the levels of FeNO. This is potentially shifting the paradigm in how investigators think of asthma management, as rising FeNO is often thought of being a bad sign. Based on this, the study investigators hypothesize that an L-citrulline-based drug strategy will normalize nitric oxide metabolism, suppress oxidative inflammatory responses and improve airway function in obese patients with asthma. The study proposal presents a clinical trial approach to treat deployment related asthma patients using L-citrulline as an add-on therapy to improve asthma control. If this confirms the investigators' previous study results, the investigators will be in route for developing the only precision-based therapy available to treat this asthma phenotype. These study results will potentially show that L-citrulline is a safe, tolerable medication that can make a significant impact on the respiratory health of a large segment of our active and veteran population at a reasonable cost.

ELIGIBILITY:
Inclusion Criteria:

* Adequate completion of informed consent process with written documentation
* Male and female patients, 18 - 70 years old, inclusive
* Meets criteria for deployment related asthma or DRA (New onset of persistent respiratory symptoms of cough, dyspnea, wheezing and/or chest tightness during or after post-9/11/2001 military deployment to Southwest Asia, accompanied by a post-bronchodilator increase in FEV1 ≥ 12% and an increase in FEV1 ≥ 200 milliliters on pulmonary function testing and/or methacholine challenge showing airways hyperresponsiveness with a 20 percent drop in FEV1 (PC[-20] FEV1) ≤ 16 mg/mL. ) Historical results from previous studies or documented in clinical records within the last 24 months are acceptable alternatives
* Able to perform reproducible spirometry according to ATS criteria
* All racial/ethnic backgrounds may participate
* Smoking tobacco history ≤15 pack years and no smoking in the last 3 months
* Suboptimal asthma control at baseline (ACQ ≥ 0.5 or ACT<19)

Exclusion Criteria:

* Respiratory tract infection within the 4 weeks prior to Visit 0
* Pulmonary-related ER visit within the 4 weeks prior to Visit 0
* Oral or systemic corticosteroid burst (for any indication) within the 4 weeks prior to Visit 0. One-time doses, such as intra-articular injections into a shoulder or knee joint, require a 2-week washout prior to Visit 0
* Significant concomitant medical illness at the discretion of the PI, including (but not limited to) heart disease, cancer, uncontrolled diabetes, other chronic lung diseases
* Chronic renal failure (creatinine > 2.0) at Visit 0 (Associated with higher ADMA levels)
* Positive urine (or serum) pregnancy test at Visit 0 or at any time during the study
* Intolerance or allergy to L-arginine or L-citrulline
* Concomitant use of PDE5 drugs or oral mononitrates
* Unable or unlikely to complete study assessments in the opinion of the Investigator
* Study intervention poses undue risk to patient in the opinion of the Investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in Asthma Control Questionnaire | Through study completion, up to 22 weeks
  To determine L-citrulline efficacy, reduction in questionnaire scores determined
Change in FeNO values | Through study completion, up to 22 weeks
  To determine L-citrulline efficacy, increase in FeNO values determined

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Holguin, MD, MPH, Principal Investigator — University of Colorado Denver- Anschutz Medical Campus
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No